CLINICAL TRIAL: NCT06802536
Title: Treatment Outcomes of Full Pulpotomy Using Two Different Calcium Silicate-based Materials in Mature Permanent Teeth With Irreversible Pulpitis Symptoms: A Randomized Clinical Trial
Brief Title: Outcomes of Full Pulpotomy Treatment in Teeth With Symptoms of Irreversible Pulpitis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Tuba Gök, PhD., Assistant Professor, Firat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIRATUNI-DENTISTRY-TUBAGOK-001
Record Dates: First submitted 2025-01-20; First posted 2025-01-31 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Pulpitis - Irreversible
Keywords: irreversible pulpitis; calcium silicate-based cement; total pulpotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Total Pulpotomy with Biodentine (Active Comparator)
  Interventions: Device: Biodentine (calcium silicate-based cement) (Septodont, Saint Maur de Fossés, France)
- Total Pulpotomy with NeoPutty (Experimental)
  Interventions: Device: NeoPutty (calcium silicate-based cement) (Avalon Biomed, Bradenton, USA)

INTERVENTIONS:
Device: Biodentine (calcium silicate-based cement) (Septodont, Saint Maur de Fossés, France) — It will be placed on the exposed pulp with the help of a carrier and the exposed pulp will be covered with material.
  Arms: Total Pulpotomy with Biodentine
Device: NeoPutty (calcium silicate-based cement) (Avalon Biomed, Bradenton, USA) — It will be placed on the exposed pulp with the help of a carrier and the exposed pulp will be covered with material.
  Arms: Total Pulpotomy with NeoPutty

SUMMARY:
The aim of this clinical trial is to learn how successful Biodentine and NeoPutty dental filling materials are in treating dental pulp inflammation in adults. It will also provide information about post-treatment pain. The main questions it aims to answer are:

Do Biodentine and NeoPutty dental filling materials treat dental pulpitis in participants? Do they reduce the need for root canal treatment?

After the application of Biodentine and NeoPutty dental filling materials to the participants, the pain and symptoms that cause pain may not decrease. In this case, the tooth may be treated with root canal treatment.

The researchers will compare the clinical success of Biodentine and NeoPutty dental filling materials with each other.

Participants will undergo a single-session pulpotomy treatment with the dental filling materials mentioned above. Clinical and radiographic follow-ups will then be performed at 3, 6 and 12 months, and records will be kept.

ELIGIBILITY:
Inclusion Criteria:

* • Patient age must be between 18-50 years

  * Must be able to give written informed consent
  * Must have systemic status (ASA 1)
  * Must have mature permanent molar or premolar (lower upper)
  * Must be symptomatic (spontaneous pain - mild to severe), extremely deep (D4) carious teeth
  * Must have pulp exposure in non-selective carious cleaning procedure
  * Must have vital response in cold test and electric pulp test
  * Must have no periodontal disease
  * Must have restorable teeth
  * Must have teeth without pulp necrosis, sinus tract or swelling/abscess
  * Must have bleeding time less than 10 minutes
  * Maximum two teeth in a patient must be included in the study (must be in different quadrants and must have at least 2 weeks between treatment periods)

Exclusion Criteria:

* Teeth with incomplete root development

  * Teeth without symptoms of irreversible pulpitis
  * Severely affected teeth that do not respond to pulp sensitivity tests
  * Teeth without signs of bleeding after exposure with the pulp chamber
  * Teeth with pulp chamber open to the oral environment
  * Teeth with periodontal pockets greater than 4 mm deep
  * Teeth with suspected cracks or crown fractures that may be responsible for pulp pathology
  * Teeth with uncontrolled bleeding
  * Medically risky patients will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-12-26 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
"Tooth survival". Both clinical and radiographic healing means "Tooth survival". Clinical healing; absence of clinical symptoms. Radiographic healing; absence of emerging periapical radiolucency. | From enrollment to the end of treatment at 1 year"

SECONDARY OUTCOMES:
"Post operative pain". It will be evaluated with a 10-unit visual analog scale. 0: no pain, 1-3 mild pain, 4-6 moderate-severe pain, 7-9 very severe pain, 10 worst pain. | From enrollment to the follow up at 1 week, 3,6.12 months"

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Title: Data Sharing for Total Pulpotomy Treatment in Teeth Diagnosed with Irreversible Pulpitis Using Biodentine and NeoPutty Materials Objective: The objective of this IPD (Individual Participant Data) sharing plan is to enhance the understanding of the success of total pulpotomy treatment in teeth diagnosed with irreversible pulpitis using Biodentine and NeoPutty materials, by encouraging and supporting data analysis.
  Data Access Conditions: Access to the data is available to researchers who present a valid proposal for research purposes and sign a data use agreement. All applications will be reviewed by the study management committee.
  Data Use: Data may only be used for scientific and ethical research purposes. Data Storage: Data will be stored for a period of ten years following the completion of the study and will be securely disposed of at the end of this period.
  Data Protection: Data will be stored under strict security protocols and accessible only to authorized personnel.
Supporting Information: Study Protocol

REFERENCES:
- [Result] European Society of Endodontology (ESE) developed by:; Duncan HF, Galler KM, Tomson PL, Simon S, El-Karim I, Kundzina R, Krastl G, Dammaschke T, Fransson H, Markvart M, Zehnder M, Bjorndal L. European Society of Endodontology position statement: Management of deep caries and the exposed pulp. Int Endod J. 2019 Jul;52(7):923-934. doi: 10.1111/iej.13080. PMID 30664240
- [Result] Duncan HF. Present status and future directions-Vital pulp treatment and pulp preservation strategies. Int Endod J. 2022 May;55 Suppl 3(Suppl 3):497-511. doi: 10.1111/iej.13688. Epub 2022 Feb 3. PMID 35080024
- [Result] Nagendrababu V, Duncan HF, Bjorndal L, Kvist T, Priya E, Jayaraman J, Pulikkotil SJ, Dummer PMH. PRIRATE 2020 guidelines for reporting randomized trials in Endodontics: explanation and elaboration. Int Endod J. 2020 Jun;53(6):774-803. doi: 10.1111/iej.13304. Epub 2020 May 9. PMID 32266988

DOCUMENTS (2):
  • Study Protocol (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT06802536/Prot_000.pdf
  • Informed Consent Form (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT06802536/ICF_001.pdf